CLINICAL TRIAL: NCT06709716
Title: Impact of Preoperative Quadratus Lumborum Block on Postoperative Opioid Consumption After Laparoscopic Hysterectomy: a Double-blinded Randomized Controlled Trial
Brief Title: Impact of Preoperative Quadratus Lumborum Block on Postoperative Opioid Consumption After Laparoscopic Hysterectomy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WRNMMC-2024-0448
Record Dates: First submitted 2024-11-15; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain; Laparoscopic Hysterectomy; Nerve Block; Quadratus Lumborum Block
Keywords: postoperative pain; quadratus lumborum block; laparoscopic hysterectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Chloride; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded parties = subject, surgical team, intraoperative anesthesia team, postoperative anesthesia team, study investigators Unblinded parties = preoperative anesthesia team (providers that perform the quadratus lumborum block)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative QL block with liposomal bupivacaine, intra-operative incisional injections with placebo (Experimental): Subjects will receive a pre-operative quadratus lumborum nerve block with liposomal bupivacaine and then an intra-operative placebo injection at each incision site with saline.
  Interventions: Drug: Quadratus Lumborum Block (QLB); Drug: Local Anesthetic Solution
- Preoperative QL block with placebo, intra-operative incisional injection with bupivacaine (Active Comparator): Subjects will undergo a sham pre-operative quadratus lumborum block procedure with saline and then an intra-operative injection of local anesthetic (0.25% bupivacaine) at each incision site.
  Interventions: Drug: Quadratus lumborum block; Drug: Local Anesthetic Solution

INTERVENTIONS:
Drug: Quadratus Lumborum Block (QLB) — Pre-operative quadratus lumborum block with liposomal bupivacaine
  Other Names: liposomal bupivacaine
  Arms: Preoperative QL block with liposomal bupivacaine, intra-operative incisional injections with placebo
Drug: Quadratus lumborum block — Pre-operative quadratus lumborum block with saline
  Other Names: saline
  Arms: Preoperative QL block with placebo, intra-operative incisional injection with bupivacaine
Drug: Local Anesthetic Solution — Intraoperative injection of 0.25% bupivacaine at each incision site
  Other Names: bupivacaine
  Arms: Preoperative QL block with placebo, intra-operative incisional injection with bupivacaine
Drug: Local Anesthetic Solution — Intraoperative injection of saline at each incision site.
  Other Names: Saline
  Arms: Preoperative QL block with liposomal bupivacaine, intra-operative incisional injections with placebo

SUMMARY:
The goal of this clinical trial is to learn if preoperative nerve block (quadratus lumborum [QL] block) works to improve pain control during and after laparoscopic hysterectomy. The main questions it aims to answer are:

Does QL block decrease the amount of narcotic medication needed during surgery? Does QL block decrease the amount of narcotic medication needed after surgery?

Researchers will compare QL block to local injection of a numbing medication at each incision site (the current standard practice) to see if QL block works to decrease surgical pain.

Participants will be randomly assigned to receive one of the two following interventions:

1. QL block before surgery with a long-acting numbing medicine (liposomal bupivacaine) and then injection of placebo (saline) at each incision site in the operating room.
2. QL block before surgery with placebo (saline) and then injection of local numbing medicine (bupivacaine) at each incision site in the operating room.

Participants will also:

* Visit the clinic/hospital for a pre-operative appointment, the surgical procedure, and a 4-6 week post-operative appointment (all standard visits even if not participating in research)
* Complete a questionnaire electronically, or by phone, that takes <10 minutes at the pre-operative appointment and on postoperative days 1, 3, 5, 14, and 4-6 weeks.

DETAILED DESCRIPTION:
Context: (Background) Given the opioid epidemic, gynecologic enhanced recovery after surgery (ERAS) pathways have been developed to reduce post-operative narcotic use through multimodal pain regimens and pre-surgical anesthetic adjuncts. While local anesthetic injection at trocar incision sites has long been accepted as a standard practice to decrease postoperative pain in laparoscopic surgery, including hysterectomy, regional nerve blockades are emerging as a promising adjunct technique for management of perioperative pain. At this time, the data evaluating the effect of regional nerve blocks on postoperative pain after laparoscopic hysterectomy are limited, thus the investigators designed the following study.

Objectives: (primary and secondary objectives) To determine the impact of preoperative quadratus lumborum (QL) block on postoperative pain following laparoscopic hysterectomy. The primary outcomes will be intraoperative and immediate post-operative opioid use, measured in morphine equivalent dose (MED). Secondary outcomes will include pain scores, functional impact of pain, perception of pain and recovery, voiding dysfunction, time to discharge, nausea/vomiting, emergency room visits, readmission, and reoperation rates.

Study Design:

This study is designed as a prospective, double-blinded, randomized controlled trial comparing opioid use in women undergoing laparoscopic hysterectomy who receive a preoperative QL block to local injection of bupivacaine (common local anesthestic).

Setting/Participants:

The study will take place at a single academic medical center that is a referral center within the military health system. Eligible patients will include adult women undergoing laparoscopic hysterectomy, including robot-assisted, that are not pain management clinic patients and don't use opioids preoperatively. Patients who have contraindications to the study protocol will be ineligible. A total of 76 patients will be enrolled with 38 in each arm.

Study Interventions and Measures:

Study arm patients will receive a preoperative bilateral QL block with an admixture of liposomal bupivacaine and 0.25% bupivacaine then an intraoperative placebo injection at each incision site with 0.9% saline. Control arm patients will receive a preoperative bilateral placebo QL block with 0.9% saline then an intraoperative injection of 0.25% bupivacaine at each incision site. Pre, intra, and postoperative care will be standardized for all study patients using the Gynecologic ERAS protocol and standard hospital perioperative procedures/protocols.

Opioid use will be measured in morphine equivalent doses (MEDs) at the intraoperative and immediate postoperative (prior to discharge) timepoints, as well as, at postoperative days 1, 3, 5, 14, and 4-6 weeks. Pain scores and impact of pain on functional status will be assessed using the DVPRS and Quality of Recovery-15 survey at these timepoints.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* scheduled to undergo laparoscopic hysterectomy
* able to speak and understand English
* DEERs eligible (eligible for healthcare within military heath system)
* Owning a phone that can receive text messages or having internet access to complete questionnaires

Exclusion Criteria:

* pre-operative opioid use
* pre-operative pain management clinic patient
* planned concomitant prolapse or incontinence procedure
* planned concomitant non-gynecologic abdominal procedure (i.e. hernia repair)
* inability to receive liposomal or non-liposomal bupivacaine
* inability to receive non-steroidal anti-inflammatory drugs (NSAIDs)
* inability to receive acetaminophen
* inability to receive oxycodone
* QL block not able to be performed bilaterally
* planned or performed mini-laparotomy (incision greater than 2cm)
* case converted to laparotomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Intraoperative opioid use | From anesthesia induction to the time the patient leaves the operating room, this is considered the "in-room time". Anticipated to be between 2-6 hours. Will be assessed up to 12 hours.
  Total opioid dose, calculated in morphine equivalent dose, required during intraoperative anesthesia care
Immediate post-operative opioid use | From time of arrival in the PACU to time of discharge from the hospital. Anticipated to be the same day, about 4-6 hours post-operative. Will be assessed up to 24 hours after surgery if the patient remains admitted.
  Total opioid dose, calculated in morphine equivalent dose, required after surgery prior to discharge from the hospital

SECONDARY OUTCOMES:
Opioid use after discharge | From discharge from the hospital to the 4-6 week post-operative appointment.
  Total opioid dose used, measured in morphine equivalent dose, from discharge to the following time points: post-operative day 1, 3, 5, 14 and 4-6 weeks post-operative.
Pain scores during inpatient post-operative care | From time of arrival in the PACU to time of discharge from the hospital. Anticipated to be the same day, about 4-6 hours post-operative. Will be assessed up to 24 hours after surgery if the patient remains admitted.
  Pain scores reported by subject in the post-operative recovery areas measured by the Defense and Veterans Pain Rating Scale (DVPRS) which ranges from 0 to 10 with 0 indicating no pain and 10 indicating pain "as bad as it can be".
Time to PACU discharge | From time of arrival in the PACU to time of transfer to the second phase of post-operative care. Anticipated to be about 1-3 hours post-operative. Will be assessed up to 12 hours after surgery if the patient remains in the PACU.
  Time from arrival to transfer out of PACU, measured in minutes
Voiding dysfunction | From time of arrival in the PACU to time of discharge from the hospital. Anticipated to be the same day, about 4-6 hours post-operative. Will be assessed up to 24 hours after surgery if the patient remains admitted.
  Inability to void post-operatively or void with inappropriately high post-void residual (urinary retention)
Pain scores after discharge | From discharge from the hospital to the 4-6 week post-operative appointment.
  Pain scores as reported by subjects on an electronic questionnaire on post-operative days 1, 3, 5, 14 and 4-6 weeks post-operative. Measured by the Defense and Veterans Pain Rating Scale (DVPRS) which ranges from 0 to 10 with 0 indicating no pain and 10 indicating pain "as bad as it can be".
Quality of Recovery-15 scores after discharge | From discharge from the hospital to the 4-6 week post-operative appointment.
  Quality of Recovery-15 scores reported by subjects by electronic questionnaire on post-operative days 1, 3, 5, 14 and 4-6 weeks post-operative. Quality of Recovery-15 scores range from 0 to 150 with higher scores indicating a better quality of recovery and lower scores indicating a poor quality of recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn A Edmonds, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edmonds K, Hunkler K, Creedon C, Drayer S, Endicott S, Eliasen K, Jones-Cox C. Impact of preoperative quadratus lumborum block on postoperative opioid consumption after laparoscopic hysterectomy: a double-blind randomized controlled trial. Pain Manag. 2025 Nov;15(11):783-790. doi: 10.1080/17581869.2025.2556648. Epub 2025 Sep 9. PMID 40923200